CLINICAL TRIAL: NCT00459745
Title: A Multi-Center, Prospective, Longitudinal, Randomized, Double-Blind, Phase III Study to Evaluate the Efficacy and Safety of Daily Administration of Pravastatin 40 mg or Fenofibrate 160 mg or Pravafen (the Combination of Pravastatin and Fenofibrate 40/160 mg) for 12 Weeks Followed by a 52-Week Open-Label Safety Phase of the Pravafen Alone in the Treatment of Combined Hyperlipidemia.
Brief Title: A Study to Evaluate Daily Pravastatin, Fenofibrate or Pravafen in the Treatment of Combined Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sc-PRAVA-06-02
Record Dates: First submitted 2007-04-09; First posted 2007-04-12 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2010-08

CONDITIONS: Combined Hyperlipidemia
Keywords: Cardiovascular Disease; Fenofibrate; LDL cholesterol; HDL cholesterol; Hyperlipidemia; Pravastatin; Triglycerides
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias | interventions — Fenofibrate; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Pravastatin (Active Comparator): Pravastatin 40 mg
  Interventions: Drug: Pravastatin
- Fenofibrate (Active Comparator): Fenofibrate 160 mg
  Interventions: Drug: Fenofibrate
- Pravafen (Parvastatin and Fenofibrate) (Experimental): Combined Therapy of Pravastatin 40 mg and Fenofibrate 160 mg.
  Interventions: Drug: Pravafen

INTERVENTIONS:
Drug: Pravafen
  Other Names: Combination of Pravastatin 40 mg and Fenofibrate 160 mg
  Arms: Pravafen (Parvastatin and Fenofibrate)
Drug: Pravastatin
  Other Names: Pravachol
  Arms: Pravastatin
Drug: Fenofibrate
  Arms: Fenofibrate

SUMMARY:
This is a multi-center, double blind, prospective, longitudinal, randomized, 12-week study with a 52-week open-label follow-up to evaluate the safety and efficacy of daily administration of Pravastatin 40 mg or Fenofibrate 160 mg or Pravafen (the combination of both Pravastatin and Fenofibrate 40/160 mg) in the treatment of combined hyperlipidemia. There will be an open-label, 8-week, Selection Phase prior to randomization in which all patients will be stabilized on Pravastatin 40 mg/day. Following the Selection Phase, and if the patients meet all inclusion/exclusion criteria, they will be randomized to a three arm, double blind, 12-week Efficacy Phase during which they would receive either Pravastatin 40 mg or Fenofibrate 160 mg or Pravafen (the combination of Pravastatin and Fenofibrate 40/160 mg). The 12-week Efficacy Phase will be followed by an open-label, 52-week, Safety Phase in which all patients will receive Pravafen.

After the 8-week Selection Phase, patients that still meet the inclusion/exclusion criteria will be randomized on a 1:1:2 ratio to Pravastatin 40 mg or Fenofibrate 160 mg or Pravafen (the combination of both Pravastatin and Fenofibrate 40/160 mg) for 12 weeks. After the completion of the 12-week double-blind phase of the study, all patients that haven't had changes in their well being, will be allowed to roll-over into the 52-week, open-label, follow-up portion of the study. During the 52 week, open label, Safety Phase of the study, all patients will receive Pravafen (the combination of Pravastatin and Fenofibrate 40/160 mg).

Patients will be evaluated at baseline and every three weeks thereafter throughout the initial 12-week Efficacy Phase of the study. Patients that roll-over into the 52-week, open-label, follow-up Safety Phase will be evaluated at 12, 24, 36 and 52 weeks.

Participation in the study can be up to 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all the criteria listed below may be selected to enroll into the Selection Phase of the study:

1. Male or female patients from 18-75 years of age, inclusive at the time of dosing with a history of a combined hyperlipidemia.
2. High LDL cholesterol and TG levels as per the table hereunder:

   Prior treatment LDL Cholesterol TG Naïve to treatment* > 130 mg/dL and ≥ 150 mg/dL and ≤ 400 mg/dL Lipid Lowering Monotherapy > 130 mg/dL and ≥ 150 mg/dL and ≤ 400 mg/dL Lipid Lowering Combination Therapy > 110 mg/dL and ≥ 150 mg/dL and ≤ 400 mg/dL

   * A patient that has received NO lipid lowering therapy within 6 weeks prior to the Selection Visit, will be considered Naïve to treatment.
3. If the patient is female and of childbearing potential and sexually active, an acceptable birth control method must be used (abstinence, IUD, oral, transdermal, injectable or implantable contraceptives, at least 2 years post-menopausal, one year post hysterectomy, double barrier device and/or partner at least one year post vasectomy), a negative serum pregnancy test must be obtained at the Selection Visit (Visit 1) and a negative urine pregnancy test must be obtained prior to study drug administration at Baseline Visit (Visit 3).
4. Able to comply with all study procedures.
5. Patients that provide a written informed consent to participate in the study indicated by a personal signature and date on the patient consent form.

At the end of the Selection Phase, patients meeting all of the criteria listed below may be selected and randomized into the Efficacy Phase of the study:

1. Selected patients with LDL Cholesterol ≥ 100 mg/dl and/or TG ≥ 150 mg/dl and ≤ 400 mg/dl at Week-1 / Visit 2 after taking Pravastatin 40 mg/day from Visit 1.
2. Patients still meeting the selection criteria a, c, d and e as listed under section 4.1.
3. Patients with a compliance ≥ 80% during the 8-week Pravastatin phase of the study.

Exclusion Criteria:

Patients will be excluded from the study if any one or more of the following apply:

1. Female of childbearing potential who is pregnant and/or lactating and/or sexually active but not using an acceptable method of contraception
2. History of allergy or contraindications to:

   * fenofibrate or similar compounds
   * HMG-CoA reductase inhibitors
3. History of uncontrolled or unstable;

   * diabetes ((i.e., diabetic nephropathy etc.),
   * hepatic impairment/insufficiency,
   * renal impairment/insufficiency (i.e., nephritis, polycystic kidney disease, acute or chronic renal failure, end-stage renal disease, GFR < 60 ml/min, etc.),
   * neurological,
   * gastrointestinal (ulcerative colitis, Barrett's, etc.),
   * gallbladder disease (patients with prior cholecystectomy can be allowed to participate),
   * psychiatric disease,
   * sleep apnea
   * any other clinically significant medical or surgical history that could affect the safety of the patient or hinder the evaluation of drug effect based on Investigator or Medical Monitor discretion
4. Acute liver disease or persistent elevations in liver function tests (2 times the upper normal limit or greater)
5. Levels of creatine phosphokinase (CK) 3 times the upper normal limit or greater
6. Change in diuretic or β-blocker treatment for hypertension within 30 days of enrollment into the selection phase (Visit 1)
7. Positive personal history of abuse of any of the following:

   * Alcohol (as per the DSM-IV criteria) and/or
   * Recreational drugs (as per the DSM-IV criteria)
8. Usage of any of the following medications (patients must have discontinued these medications for 5 or more half-lives or for 30 days, whichever is greater prior to study drug administration on Visit 3 / Day 0) :

   * Corticosteroids
   * Immunosuppressants
   * Macrolide antibiotics
   * Azole antifungal agents, or
9. Recent use of any investigational drug. These drugs must have been discontinued for either 5 or more half-lives or for 30 days whichever is greater prior to Visit 1
10. Hyperlipidemia type I-IIa-IV-V
11. LDL < 100 mg/dL
12. TG < 150 mg/dL or > 400 mg/dL
13. Uncontrolled primary hypothyroidism
14. History of an acute myocardial infarction, stroke within the last 6 month prior to Visit 1; unstable angina or clinically significant heart failure
15. Uncontrolled hypertension, as defined by SBP >160 mmHg or DBP >100 mmHg while on anti-hypertensive medication
16. Type 1 diabetes or type 2 diabetes mellitus requiring insulin, and diabetic patients with poor control (HbA1c level > 8.5%), abnormal renal function (GFR < 60 ml/mn) or any renal disease likely to lead to renal dysfunctions)
17. Use of any of the prohibited medications as detailed in the concomitant medication section
18. Non adherence to the American Heart Association Step II diet introduced at Visit 1
19. Presence of any other condition or illness, which, in the opinion of the Principal Investigator, would interfere with the patient's participation in the study

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Primary endpoints will assess differences in change from baseline in non-HDL-C, for the patients receiving Pravafen versus the patients receiving Pravastatin or Fenofibrate at the end of the 12-week portion of the study. | bBaseline to 12 weeks
  Change in HDL

SECONDARY OUTCOMES:
Secondary endpoints will assess differences in change from baseline in TC, TG, LDL-C, HDL-C and TC/HDL-C for the pts receiving the combo therapy vs the pts receiving Pravastatin or Fenofibrate | Baseline to 12 weeks
  Changes in TC, TG, LDL-C, HDL-C and TC/HDL-C
Differences in change from baseline in ALT, AST and CK as well as overall safety for the pts receiving the combo therapy vs the pts receiving Pravastatin or Fenofibrate at the end of the 12-week of the study | Baseline to 12 weeks
  Changes in ALT, AST and CK and overall safety

CONTACTS AND LOCATIONS:
Locations (56):
- United States (56):
  - Anasazi Internal Medicine, Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Memorial Research Medical Clinic, Long Beach, California
  - Clinical Trials Research, Roseville, California
  - Orange County Research Center, Tustin, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Drug Study Institute, Jupiter, Florida
  - Mima Century Research Associates, Melbourne, Florida
  - Cardiology Research Associates, Ormond Beach, Florida
  - Atlanta Vascular Research Foundation, Atlanta, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Welborn Clinic Research Center, Evansville, Indiana
  - MediSphere Medical Research Center LLC, Evansville, Indiana
  - Research Institute of Middle America, Jeffersonville, Indiana
  - Welborn Clinic Gateway, Newburgh, Indiana
  - Lemarc Research Center, Louisville, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Androscoggin Cardiology Associates, Auburn, Maine
  - MODEL Clinical Research, Baltimore, Maryland
  - Health Trends Research, LLC, Baltimore, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Clinical Research Center of Cape Cod, Inc, West Yarmouth, Massachusetts
  - Clinical Study Site, Florissant, Missouri
  - Mercy Medical Group, Manchester, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Bronx Nephrology Hypertension, P.C., The Bronx, New York
  - Capital Cardiology Associates, Troy, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Sensenbrenner Primary Care LLC, Charlotte, North Carolina
  - Triangle Medical Research Associates, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Crescent Medical Research Associates, Salisbury, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Sterling Research Group, Cincinnati, Ohio
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Ohio Clinical Research, Hudson, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Ohio Clinical Research, LLC, Lyndhurst, Ohio
  - Bluestem Cardiology, Bartlesville, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Southern Berks Family Medicine, Reading, Pennsylvania
  - Tipton Medical Center, Tipton, Pennsylvania
  - Palmetto Medical Research Associates, Mt. Pleasant, South Carolina
  - Upstate Pharmaceutical Research, Simpsonville, South Carolina
  - TriCities Medical Research Associates, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Trials Research, Austin, Texas
  - Texas Medical Research LLC, San Antonio, Texas
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - National Clinical Research, Richmond, Virginia
  - Rainier Clinical Research Center Inc., Renton, Washington
  - Cedar Research LLC, Tacoma, Washington